Randomized Controlled Trial of Inferior Vena Cava Ultrasonography in the Management and Disposition of Pediatric Patients Undergoing Evaluation for Sepsis and Dehydration

PI: Dr. James Tsung NCT02568189

Document Date: 05-08-2015


Study ID #: IF1733382 Form Version Date:05/08/2015

#### TITLE OF RESEARCH STUDY:

Title: Utility of Inferior Vena Cava Ultrasonography in the Management and Disposition of Pediatric Patients Undergoing Evaluation for Sepsis and Dehydration

#### PRINCIPAL INVESTIGATOR (HEAD RESEARCHER) NAME AND CONTACT INFORMATION:

Name: Elizabeth Haines DO

Physical Address: Emergency Department, Guggenheim Pavilion, Main Corridor

Mailing Address: 1 Gustave L Levy Place Box 1149, NY, NY 10029

Phone: 212-241-6272

## WHAT IS A RESEARCH STUDY?

A research study is when scientists try to answer a question about something that we don't know enough about. Participating may not help you or others.

People volunteer to be in a research study. The decision about whether or not to take part is totally up to you. You can also agree to take part now and later change your mind. Whatever you decide is okay. It will not affect your ability to get medical care within the Mount Sinai Health System.

Someone will explain this research study to you. Feel free to ask all the questions you want before you decide. Any new information that develops during this research study that might make you change your mind about participating will be given to you promptly.

Basic information about this study will appear on the website http://www.ClinicalTrials.gov. There are a few reasons for this: the National Institutes of Health (NIH) encourages all researchers to post their research; some medical journals only accept articles if the research was posted on the website; and, for research studies the U.S. Food and Drug Administration (FDA) calls "applicable clinical trials" a description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

### **PURPOSE OF THIS RESEARCH STUDY:**

The purpose of this study is to use point-of-care (bedside) ultrasound, which is an experimental technique, to look at your inferior vena cava (large vein bringing blood to the heart) to see if the size of the inferior vena cava (flat versus normal for age or plump) changes the way we treat your condition. With the information obtained from your ultrasound, researchers will see if medical treatments which may have been used later within the ER visit where given sooner and if it decreases the ER length of stay among all research participants.

# This Section For IRB Official Use Only This Consent Document is approved for use by an Institutional Review Board (IRB) Form Approval Date: DO NOT SIGN AFTER THIS DATE →

Rev. 4/1/15 IRB Form HRP-502a

# THE MOUNT SINAI HEALTH SYSTEM CONSENT FORM TO VOLUNTEER IN A RESEARCH STUDY AND AUTHORIZATION FOR USE AND DISCLOSURE OF MEDICAL INFORMATION

Icahn School of Medicine at Mount Sinai,

### 

## Study ID #: IF1733382

Form Version Date: 05/08/2015

You may qualify to take part in this research study because you are exhibiting signs of a serious bacterial or viral infection causing sepsis (whole-body inflammation caused by an infection) or dehydration (loss of more fluid than taken in) from vomiting and/or diarrhea.

Funds for conducting this research are provided by Mount Sinai

# LENGTH OF TIME AND NUMBER OF PEOPLE EXPECTED TO PARTICIPATE

Your participation in this research study is expected to last for the length of the ER visit.

The number of people expected to take part in this research study at the Ichan School of Medicine at Mount Sinai is 564 participants.

# **DESCRIPTION OF WHAT'S INVOLVED:**

If you agree to participate in this research study, the following information describes what may be involved.

If you agree to participate in this research study, the following information describes what may be involved.

- Once you consent to enroll in this study, you will be assigned randomly to one of two groups. The
  group to which you will be assigned will be chosen by chance, like flipping a coin. Neither you nor
  the study doctor will choose what study treatment you get. You will have an equal chance of being
  given each study treatment.
- One group will have an ultrasound of the inferior vena cava before any tests or treatment is given
  to you. Inferior vena cava ultrasound is an investigational technique, whose role in the
  management of sepsis and dehydration has not yet been established. The aim of this study is to
  see if inferior vena cava ultrasound will be able to change the way we treat your condition.
- The other group will have an inferior vena cava ultrasound performed 15 minutes after receiving IV fluids or fluids by mouth. As noted above, inferior vena cava ultrasound is an investigational technique, whose role in the management of sepsis and dehydration has not yet been established. The aim of this study is to see if inferior vena cava ultrasound will be able to change the way we treat your condition.
- An inferior vena cava ultrasound is like having a video of the inside of the abdomen. The doctor
  will use a small, smooth probe coated with a thin layer of jelly and place it on your abdomen. This
  test is also pain-free and will take approximately 3-5 minutes. There is zero radiation exposure
  with all ultrasound studies.

If you agree to participation in this research study, the ER staff will document the results of the inferior vena cava ultrasound as well as collect other relevant information including your vital signs such as temperature, heart rate, respiratory rate (breathing rate), and oxygen saturation, and medical treatment that was given in the ER as a result of the ultrasound.

# This Section For IRB Official Use Only

| This Consent Document is approved for use by an Institutional Review Board (IRB) | | |
|---|---|---|
| Form Approval Date: | DO NOT SIGN AFTER THIS DATE $ ightarrow$ | |
| Rev. 4/1/15 | • | IRB Form HRP-502a |


Study ID #: IF1733382

Form Version Date: 05/08/2015

#### YOUR RESPONSIBILITIES IF YOU TAKE PART IN THIS RESEARCH:

If you decide to take part in this research study you will be responsible for the following things:

- Consenting to take part in this research study
- Participating with the ultrasound in the E.R.
- Following your E.R. doctor's discharge instructions.

## COSTS OR PAYMENTS THAT MAY RESULT FROM PARTICIPATION:

You will not be paid for participating in this research study. Being in this research study will not lead to extra costs to you. You will not be reimbursed for your travel or time that may be required for study visits.

# **POSSIBLE BENEFITS:**

It is important to know that you may not get any benefit from taking part in this research. Others may not benefit either. However, your participation in this study may lead to getting necessary medical interventions sooner because of the findings of the inferior vena cava ultrasound.

#### REASONABLY FORESEEABLE RISKS AND DISCOMFORTS:

There may be slight discomfort from contact with ultrasound gel and probe on the abdomen. If you experience discomfort the exam will be discontinued. In previous similar research studies, no one reported any discomfort from the ultrasound examination.

There always exists the potential for loss of private information; however, there are procedures in place to minimize this risk.

#### OTHER POSSIBLE OPTIONS TO CONSIDER:

You may decide not to take part in this research study without any penalty. The choice is totally up to you. Instead of being in this research study, you may choose to proceed with the routine, standard of care treatments for suspected sepsis or dehydration recommended by your E.R. doctor.

#### IN CASE OF INJURY DURING THIS RESEARCH STUDY:

If you believe that you have suffered an injury related to this research as a participant in this study, you should contact the Principal Investigator at (212) 241-6272.

| This Section For IRB Official Use Only | | | |
|---|---|---|---|
| This Consent Document is approved for use by an Institutional Review Board (IRB) | | | |
| Form Approval Date: | DO NOT SIGI | N AFTER THIS DATE → | |
| Rev. 4/1/15 | | | IRB Form HRP-502a |


Study ID #: IF1733382 Form Version Date:05/08/2015

#### ENDING PARTICIPATION IN THE RESEARCH STUDY:

You may stop taking part in this research study at any time without any penalty. This will not affect your ability to receive medical care at any of the Mount Sinai Health System hospitals or to receive any benefits to which you are otherwise entitled.

If you decide to stop being in the research study, please contact the Principal Investigator or the research staff.

You may also withdraw your permission for the use and disclosure of any of your protected information for research, but <u>you must do so in writing</u> to the Principal Investigator at the address on the first page. Even if you withdraw your permission, the Principal Investigator for the research study may still use the information that was already collected if that information is necessary to complete the research study. Your health information may still be used or shared after you withdraw your authorization if you have an adverse event (a bad effect) from participating in the research study.

<u>Withdrawal without your consent</u>: The study doctor, the sponsor or the institution may stop your involvement in this research study at any time without your consent. This may be because the research study is being stopped, the instructions of the study team have not been followed, the investigator believes it is in your best interest, or for any other reason. If specimens or data have been stored as part of the research study, they too can be destroyed without your consent.

# **CONTACT PERSON(S):**

If you have any questions, concerns, or complaints at any time about this research, or you think the research has hurt you, please contact the office of the research team and/or the Principal Investigator at phone number (212) 241-6272 (office) or (516) 946-9742 (mobile).

This research has been reviewed and approved by an Institutional Review Board. You may reach a representative of the Program for Protection of Human Subjects at the Icahn School of Medicine at Mount Sinai at telephone number (212) 824-8200 during standard work hours for any of the reasons listed below. This office will direct your call to the right person within the Mount Sinai Health System:

- Your questions, concerns, or complaints are not being answered by the research team.
- You cannot reach the research team.
- You are not comfortable talking to the research team.
- You have questions about your rights as a research subject.
- You want to get information or provide input about this research.

# **DISCLOSURE OF FINANCIAL INTERESTS:**

Sometimes, physicians/researchers receive payments for consulting or similar work performed for industry. Effective September 2014 Mount Sinai reviews only payments to an individual totaling more than \$5,000 a year per entity when determining potential conflicts of interest. If you have questions

#### This Section For IRB Official Use Only

| This Consent Document is approved for use by an Institutional Review Board (IRB) | | |
|---|---|---|
| Form Approval Date: | DO NOT SIGN AFTER TI | HIS DATE → |
| Rev. 4/1/15 | | IRB Form HRP-502a |

# THE MOUNT SINAI HEALTH SYSTEM CONSENT FORM TO VOLUNTEER IN A RESEARCH STUDY AND AUTHORIZATION FOR USE AND DISCLOSURE OF MEDICAL INFORMATION

Icahn School of Medicine at Mount Sinai,

### 

## Study ID #: IF1733382

Form Version Date: 05/08/2015

regarding industry relationships, we encourage you to talk your physician/researcher or visit our website at http://icahn.mssm.edu/ where Mount Sinai publicly discloses the industry relationships of our faculty.

#### **MAINTAINING CONFIDENTIALITY - HIPAA AUTHORIZATION:**

As you take part in this research project it will be necessary for the research team and others to use and share some of your private protected health information. Consistent with the federal Health Insurance Portability and Accountability Act (HIPAA), we are asking your permission to receive, use and share that information.

What protected health information is collected and used in this study, and might also be disclosed (shared) with others?

As part of this research project, the research team at the hospital(s) involved in the research will collect your name, telephone number, medical record number, date of birth, radiographic data, admission date.

The researchers will also get information from your medical record from the Ichan School of Medicine at Mount Sinai.

During the study the researchers will gather information by:

- taking a medical history (includes current and past medications or therapies, illnesses, conditions or symptoms, family medical history, allergies, etc.)
- doing a physical examination that generally also includes blood pressure reading, heart rate, breathing rate and temperature
- completing the tests, procedures, questionnaires and interviews explained in the description section of this consent.

#### Why is your protected health information being used?

Your health information and the results of any tests and procedures being collected as part of this research study will be used for the purpose of this study as explained earlier in this consent form. The results of this study could be published or presented at scientific meetings, lectures, or other events, but would not include any information that would let others know who you are, unless you give separate permission to do so.

The research team and other authorized members of The Mount Sinai Health System ("Mount Sinai") workforce may use and share your information to ensure that the research meets legal, institutional or accreditation requirements. For example, the School's Program for the Protection of Human Subjects is responsible for overseeing research on human subjects, and may need to see your information. If you receive any payments for taking part in this study, the Mount Sinai Finance Department may need your name, address, social security number, payment amount, and related information for tax reporting purposes. If the research team uncovers abuse, neglect, or reportable diseases, this information may be disclosed to appropriate authorities.

# This Section For IRB Official Use Only

| This Consent Document is approved for use by an Institutional Review Board (IRB) | | |
|---|---|---|
| Form Approval Date: | DO NOT SIGN AFTER THIS DATE $\rightarrow$ | |
| Rev. 4/1/15 | • | IRB Form HRP-502a |


#### Study ID #: IF1733382

Form Version Date:05/08/2015

Who, outside Mount Sinai, might receive your protected health information?

As part of the study, the Principal Investigator, study team and others in the Mount Sinai workforce may disclose your protected health information, including the results of the research study tests and procedures, to the following people or organizations: (It is possible that there may be changes to the list during this research study; you may request an up-to-date list at any time by contacting the Principal Investigator.)

- A Data Safety Monitoring Board or other committee that will monitor the study on an ongoing basis for safety.
- The United States Department of Health and Human Services and the Office of Human Research Protection.

In all disclosures outside of Mount Sinai, you will not be identified by name, social security number, address, telephone number, or any other direct personal identifier unless disclosure of the direct identifier is required by law. Some records and information disclosed may be identified with a unique code number. The Principal Investigator will ensure that the key to the code will be kept in a locked file, or will be securely stored electronically. The code will not be used to link the information back to you without your permission, unless the law requires it, or rarely if the Institutional Review Board allows it after determining that there would be minimal risk to your privacy. It is possible that a sponsor or their representatives, a data coordinating office, a contract research organization, may come to inspect your records. Even if those records are identifiable when inspected, the information leaving the institution will be stripped of direct identifiers. Additionally, when applicable, the monitors, auditors, the IRB, the Office of Human Subjects Protection (OHRP) of the Department of Health and Human Services as well as the Food and Drug Administration (FDA) will be granted direct access to your medical records for verification of the research procedures and data. OHRP and FDA are authorized to remove information with identifiers if necessary to complete their task. By signing this document you are authorizing this access. We may publish the results of this research. However, we will keep your name and other identifying information confidential.

For how long will Mount Sinai be able to use or disclose your protected health information? Your authorization for use of your protected health information for this specific study does not expire.

### Will you be able to access your records?

During your participation in this study, you will not be able to access your medical records. This will be done to prevent the knowledge of study results from affecting the reliability of the study. Your information will be available should an emergency arise that would require your treating physician to know this information to best treat you. You will have access to your medical record and any study information that is part of that record when the study is over or earlier, if possible. The investigator is not required to release to you research information that is not part of your medical record.

### Do you need to give us permission to obtain, use or share your health information?

NO! If you decide not to let us obtain, use or share your health information you should not sign this form, and you will not be allowed to volunteer in the research study. If you do not sign, it will not affect your treatment, payment or enrollment in any health plans or affect your eligibility for benefits.

| This Section For IRB Official Use Only | | |
|---|---|---|
| This Consent Document is approved for use by an Institutional Review Board (IRB) | | |
| Form Approval Date: | DO NOT SIGN AFTER THIS DATE $\rightarrow$ | |
| Rev. 4/1/15 | | IRB Form HRP-502a |


Study ID #: IF1733382 Can you change your mind? Form Version Date: 05/08/2015

You may withdraw your permission for the use and disclosure of any of your protected information for research, but you must do so in writing to the Principal Investigator at the address on the first page. Even if you withdraw your permission, the Principal Investigator for the research study may still use your protected information that was already collected if that information is necessary to complete the study. Your health information may still be used or shared after you withdraw your authorization if you should have an adverse event (a bad effect) from being in the study. If you withdraw your permission to use your protected health information for research that means you will also be withdrawn from the research study, but standard medical care and any other benefits to which you are entitled will not be affected. You can also tell us you want to withdraw from the research study at any time without canceling the Authorization to use your data.

It is important for you to understand that once information is disclosed to others outside Mount Sinai, the information may be re-disclosed and will no longer be covered by the federal privacy protection regulations. However, even if your information will no longer be protected by federal regulations, where possible, Mount Sinai has entered into agreements with those who will receive your information to continue to protect your confidentiality.

If as part of this research project your medical records are being reviewed, or a medical history is being taken, it is possible that HIV-related information may be revealed to the researchers. If that is the case, the following information concerns you. If this research does not involve any review of medical records or questions about your medical history or conditions, then the following section may be ignored.

#### **Notice Concerning HIV-Related Information**

If you are authorizing the release of HIV-related information, you should be aware that the recipient(s) is (are) prohibited from re-disclosing any HIV-related information without your authorization unless permitted to do so under federal or state law. You also have a right to request a list of people who may receive or use your HIV-related information without authorization. If you experience discrimination because of the release or disclosure of HIV-related information, you may contact the New York State Division of Human Rights at (888) 392-3644 or the New York City Commission on Human Rights at (212) 306-5070. These agencies are responsible for protecting your rights.

[Omit the signature page if there is no written documentation of consent.]

| This Section For IRB Official Use Only | | |
|---|---|---|
| This Consent Document is approved for use by an Institutional Review Board (IRB) | | |
| Form Approval Date: | DO NOT SIGN AFTER THIS DATE $\rightarrow$ | |
| Rev. 4/1/15 | • | IRB Form HRP-502a |

# THE MOUNT SINAI HEALTH SYSTEM CONSENT FORM TO VOLUNTEER IN A RESEARCH STUDY AND AUTHORIZATION FOR USE AND DISCLOSURE OF MEDICAL INFORMATION

Icahn School of Medicine at Mount Sinai,


Form Version Date:05/08/2015 Study ID #: IF1733382 Signature Block for Capable Adult Your signature below documents your permission to take part in this research and to the use and disclosure of your protected health information. A signed and dated copy will be given to you. DO NOT SIGN THIS FORM AFTER THIS DATE Signature of subject Date Printed name of subject Time frequired if used for FDA documentation purposes] Person Explaining Study and Obtaining Consent Signature of person obtaining consent Date Printed name of person obtaining consent Time Witness Section: For use when a witness is required to observe the consent process,, document below (for example, subject is illiterate or visually impaired, or this accompanies a short form consent): My signature below documents that the information in the consent document and any other written information was accurately explained to, and apparently understood by, the subject, and that consent was freely given by the subject. Signature of witness to consent process Date Printed name of person witnessing consent process Time This Section For IRB Official Use Only This Consent Document is approved for use by an Institutional Review Board (IRB) DO NOT SIGN AFTER THIS DATE → Form Approval Date:

Rev. 4/1/15 IRB Form HRP-502a